CLINICAL TRIAL: NCT07089693
Title: Determination of Risk Factors, Incidence and Mortality Rates of Acute Kidney Injury in COVID-19 Patients Hospitalized in Intensive Care Unit
Brief Title: Acute Kidney Injury in Critical COVID-19: Outcomes and Risks
Status: Completed | Type: Observational
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Pınar KARABAK BİLAL, MD, Intensive Care Specialist, Ankara University
Other Study IDs: İ05-257-22
Record Dates: First submitted 2025-07-21; First posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: COVID -19; Acute Kidney Injury; Intensive Care Unit (ICU) Admission; Mortality
Keywords: COVID-19; acute kidney injury; intensive care unit; risk factors; incidence
MeSH Terms: conditions — COVID-19; Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- non-AKI
- stage 1 AKI
- stage 2 AKI
- stage 3 AKI

SUMMARY:
This retrospective observational study aims to determine the incidence of acute kidney injury (AKI) associated with COVID-19, risk factors, and effects on mortality for intensive care unit patients. Data from 238 COVID-19 patients monitored in the Anesthesiology and Reanimation Intensive Care Unit of Ankara University Ibni Sina Hospital between January 1, 2021 and January 1, 2022 were retrospectively reviewed. Patients were divided into two groups according to the level of renal damage (with and without AKI). Those with AKI were staged per the KDIGO criteria (Stage 1-2-3). Demographic data, comorbidities, Charlson comorbidity indexes, Acute Physiology and Chronic Health Evaluation scores, laboratory results, and mortality data were examined. The data obtained were compared between the groups.

The findings may help improve clinical awareness and guide management strategies in intensive care unit patients with COVID-19 at risk of AKI

DETAILED DESCRIPTION:
This retrospective, single-center observational study was conducted at Ankara University Hospital. Data from 238 COVID-19 patients monitored in the Anesthesiology and Reanimation Intensive Care Unit of Ankara University Ibni Sina Hospital between January 1, 2021 and January 1, 2022 were retrospectively reviewed. The objective of the study was to investigate the frequency, risk factors, and impact on mortality of acute kidney injury (AKI) in adult patients hospitalized with confirmed COVID-19 infection.

Patients with a confirmed diagnosis of COVID-19 and available renal function data were included in the analysis. AKI was defined and staged according to the Kidney Disease: Improving Global Outcomes (KDIGO) criteria. Demographic characteristics, comorbidities, laboratory values, and clinical parameters were evaluated to identify potential risk factors for AKI development. The relationship between the presence and severity of AKI and in-hospital mortality was assessed.

The study aims to provide insight into the burden of COVID-19-associated AKI and to support improved clinical decision-making for identifying and managing high-risk patients in hospital settings.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Hospitalized patients with COVID-19 confirmed by PCR test
* Required follow-up in the intensive care unit between January 1, 2021 and January 1, 2022

Exclusion Criteria:

* Patients with end-stage renal disease (ESRD)
* History of renal transplantation
* Intensive care unit stay shorter than 48 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (aged 18 and older) with PCR-confirmed COVID-19 who were admitted to the intensive care unit (ICU) at Ankara University Hospital between January 1,2021 and January 1,2022. All patients had available records and remained in the ICU for at least 48 hours.
Sampling Method: Non-Probability Sample
Enrollment: 238 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-08-15 (Actual)

PRIMARY OUTCOMES:
Intensive care unit mortality | From ICU admission until in-hospital death or ICU discharge, whichever occurs first, assessed up to 90 days.
  To evaluate whether the development of AKI is associated with mortality in COVID-19 patients monitored in the intensive care unit.

SECONDARY OUTCOMES:
Length of intensive care unit stay | From ICU admission until ICU discharge, assessed up to 12 months.
  To assess whether the development of AKI in COVID-19 patients is associated with the length of stay in the intensive care unit.
Incidence of acute kidney injury | From ICU admission until AKI diagnosis or ICU discharge, whichever occurs first, assessed during hospitalization (up to 100 days).
  To determine the incidence of AKI among COVID-19 patients, defined by the KDIGO criteria.
Association between patient characteristics and AKI development | From ICU admission until AKI diagnosis or ICU discharge, assessed up to 100 days.
  To identify clinical and laboratory predictors associated with AKI development in COVID-19 patients requiring intensive care, using retrospective data analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Gizem Kahraman, MD, Principal Investigator — Ankara University Department of Anesthesiology and Reanimation; Mustafa Kemal Bayar, Prof, Study Director — Ankara University Department of Anesthesiology and Reanimation; Pınar Karabak Bilal, MD, Principal Investigator — Ankara University Department of Anesthesiology and Reanimation
Locations (1):
- Ankara University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arentz M, Yim E, Klaff L, Lokhandwala S, Riedo FX, Chong M, Lee M. Characteristics and Outcomes of 21 Critically Ill Patients With COVID-19 in Washington State. JAMA. 2020 Apr 28;323(16):1612-1614. doi: 10.1001/jama.2020.4326. PMID 32191259
- [Background] Ratnayake A, Sarnowski A, Sinclair F, Annear NMP, Banerjee D, Chis Ster I. The dynamics and outcomes of AKI progression during the COVID-19 pandemic. Nephrology (Carlton). 2024 Jun;29(6):325-337. doi: 10.1111/nep.14297. Epub 2024 Mar 28. PMID 38549280
- [Background] Guissouma J, Ben Ali H, Allouche H, Trabelsi I, Hammami O, Yahia Y, Hatem G. Acute Kidney Injury Complicating Critical Forms of COVID-19: risk Factors and Prognostic Impact. F1000Res. 2025 Jan 2;13:497. doi: 10.12688/f1000research.144105.3. eCollection 2024. PMID 39839732
- [Background] Aklilu AM, Kumar S, Nugent J, Yamamoto Y, Coronel-Moreno C, Kadhim B, Faulkner SC, O'Connor KD, Yasmin F, Greenberg JH, Moledina DG, Testani JM, Wilson FP. COVID-19-Associated Acute Kidney Injury and Longitudinal Kidney Outcomes. JAMA Intern Med. 2024 Apr 1;184(4):414-423. doi: 10.1001/jamainternmed.2023.8225. PMID 38407862